CLINICAL TRIAL: NCT02355002
Title: Transcranial Magnetic Stimulation (TMS) in Obsessive Compulsive Disorder (OCD): Mechanisms and Biomarkers
Acronym: TMSOCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Joan A Camprodon, MD MPH PhD, MD, MPH, PhD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2014P002560
Record Dates: First submitted 2015-01-30; First posted 2015-02-04 (Estimated); Results first posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-05

CONDITIONS: Obsessive Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active Transcranial Magnetic Stimulation (TMS) treatment (Experimental): In this arm subjects will receive real, active TMS with a standard, water-cooled, figure-8 shaped TMS coil.
  Interventions: Device: Transcranial Magnetic Stimulation
- Sham-TMS treatment (Sham Comparator): This arm serves as the sham/placebo control. In TMS a sham coil is used to create a sensory experience which is similar to active TMS, but in which the magnetic field is blocked by a metal shield built into the coil.
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Transcranial magnetic stimulation uses a rapidly changing magnetic field to induce current in brain tissue non-invasively. It is common procedure in both clinical and research settings, and it has well established guidelines for safe an ethical use which maximize safety for all subjects.

SUMMARY:
The purpose of this study is to test the efficacy of 1-Hz repetitive transcranial magnetic stimulation (TMS) over the pre-supplementary motor area as a treatment for obsessive compulsive disorder. Additionally, this study aims to identify the mechanisms of action of TMS and potential biomarkers and predictors of treatment response.

DETAILED DESCRIPTION:
This treatment study examines the use of transcranial magnetic stimulation (TMS) in treating people with OCD and investigates what areas of the brain are involved during emotional learning. TMS is a noninvasive method in which a magnetic "coil" is placed near an individual's head and delivers small magnetic pulses into the brain, which produce small electrical currents in the brain, stimulating brain cells that may relieve OCD symptoms. TMS has been FDA approved since 2008 and Health Canada approved since 2002 as a treatment for depression. Our hope is to demonstrate that TMS is a successful treatment option for individuals struggling with OCD symptoms, and to identify the specific areas of the brain that are targeted through TMS.

Patients will be randomized (like the flip of a coin) to one of two groups: 6 weeks of daily active TMS, or 6 weeks of daily placebo (sham) TMS sessions. During phase I, participation in this study will last about 8 weeks and patients will be asked to make about 36 visits to our clinics at the MGH main campus and the MGH Charlestown Navy Yard campus. Patients will also participate in MRI scanning sessions and clinical assessments.

If patients' symptoms do not improve after phase I, they will be invited to participate in phase II. During phase II, patients receive 30 active TMS sessions over 6 weeks, as well as MRI scans and clinical assessments.

Part of the MRI scanning sessions will include participating in a task that uses mild, half-second electric shocks to fingers. The electric current will be generated from a 9V battery (e.g., battery in a smoke alarm), and is much less annoying than a static shock. In order to set the level of the current to be used during the study, we will begin at a level below what patients will be able to feel, and then increase in gradual steps with permission. Patients will be asked to stop the increase at a level of the current that they find highly annoying but not painful. The level of current that patients select during this trial procedure, and no higher level, will be used during the study so that they will not receive any painful electric shocks. The purpose of the electric shock is to create a situation in which emotional learning may occur. Patients will receive no more than ten of these electric shocks.

Compensation is provided for clinical assessments and MRI scan sessions.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years of age.
2. Proficient in English.
3. A diagnosis of primary OCD (as determined by SCID).
4. Yale-Brown Obsessive Compulsive Scale total score ≥ 16.
5. Normal (or corrected) vision.
6. Stable medication regimen or medication free for ≥ 12 weeks prior to study; benzodiazepine free ≥ 2 weeks.
7. Right-handed (Edinburgh Handedness Inventory - Short Form total score ≥ 61)
8. Able to give informed consent.

Exclusion Criteria:

1. Current or history of neurologic or psychiatric disease (e.g., mental retardation, dementia, brain damage, or other cognitive impairment) that would interfere with ability to engage in TMS
2. Psychopathology not appropriate for the treatment (e.g., manic episode or psychosis)
3. Substance abuse or dependence that is current or within the last six months or use of an illicit drug that is not prescribed, as indicated by a urine drug screen and/or clinical inference.
4. Use of benzodiazepines or anticonvulsants within 2 weeks prior to study (to be ruled out by a urine drug screen).
5. Use of Tricyclic Antidepressants (e.g. Clomipramine).
6. Use of other psychotropic medications (e.g., SSRIs) will be allowed provided the dose has been stable for > 12 weeks.
7. Documented resistance to 4 or more valid pharmacological trials of 2 or more different medication classes (e.g. SSRIs and TCAs).
8. Previous exposure to TMS.
9. Major/chronic medical conditions.
10. History of head injury resulting in prolonged loss of consciousness and/or neurological sequelae.
11. Prior neurosurgical procedure.
12. Metal in the body, metal injury to the eyes.
13. History of seizures.
14. Implanted pacemaker, medication pump, vagal stimulator, deep brain stimulator, TENS unit, or ventriculo-peritoneal shunt
15. Pregnancy; breastfeeding or nursing; for women of childbearing a pregnancy test (to be ruled out by urine β-HCG) will be conducted prior to study.
16. Currently in Cognitive Behavioral Therapy (CBT).
17. Diagnosis of primary sleep disorder such as primary insomnia, narcolepsy, sleep apnea, shift work sleep disorder and others. Sleep disorders such as insomnia or hypersomnia that are secondary to depression or OCD are permitted.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-05; Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joan A Camprodon, MD, MPH, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Transcranial Magnetic Stimulation (TMS) Treatment: In this arm subjects will receive real, active TMS with a standard, water-cooled, figure-8 shaped TMS coil.
  Transcranial Magnetic Stimulation: Transcranial magnetic stimulation uses a rapidly changing magnetic field to induce current in brain tissue non-invasively. It is common procedure in both clinical and research settings, and it has well established guidelines for safe an ethical use which maximize safety for all subjects. See attached Rossi et. al. 2009 as a reference to safety guidelines for TMS.
- Sham-TMS Treatment: This arm serves as the sham/placebo control. In TMS a sham coil is used to create a sensory experience which is similar to active TMS, but in which the magnetic field is blocked by a metal shield built into the coil.
  Transcranial Magnetic Stimulation: Transcranial magnetic stimulation uses a rapidly changing magnetic field to induce current in brain tissue non-invasively. It is common procedure in both clinical and research settings, and it has well established guidelines for safe an ethical use which maximize safety for all subjects. See attached Rossi et. al. 2009 as a reference to safety guidelines for TMS.
Period: Period 1: Phase 1, Randomized-Controlled
Arm/Group | Active Transcranial Magnetic Stimulation (TMS) Treatment | Sham-TMS Treatment
Started | 15 | 11
Completed | 12 | 10
Not Completed | 3 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawn by principal investigator due to start of the COVID-19 lock-down | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Period: Period 2: Phase 2 Open-Label
Arm/Group | Active Transcranial Magnetic Stimulation (TMS) Treatment | Sham-TMS Treatment
Started (Six participants from the phase I RCT (2 active TMS, 4 sham) showed sufficient symptom improvement and were not invited to participate in the phase II open-label treatment. All other phase I completers were invited to receive open-label, active TMS in phase II (there were no sham participants in phase II).) | 16 | 0
Completed | 12 | 0
Not Completed | 4 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Participant left country | 1 | 0
Not completed — Withdrawn by principal investigator due to start of the COVID-19 lock-down | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Transcranial Magnetic Stimulation (TMS) Treatment | Sham-TMS Treatment | Total
Number analyzed (Participants) | 15 | 11 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 11 | 26
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 6 | 6 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 7 | 20
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 15 | 11 | 26

OUTCOME MEASURES:

1. Primary Outcome: Obsessive Compulsive Symptoms as Measured by Yale-Brown Obsessive Compulsive Scale (Y-BOCS)
Description: The Yale-Brown Obsessive Compulsive Scale (Y-BOCS) is the gold-standard, semi-structured clinician-administered assessment of OCD symptom severity. It contains 10 items ranging from 0 (no symptoms) to 4 (extreme symptoms), yielding a total possible score range from 0 to 40. Higher scores indicate more severe OCD symptom severity. We compared the efficacy of TMS to Sham in reducing OCD symptom severity over a 6-week period. Efficacy was again compared in the follow-up phase of the study in from week 6 to week 18.
Time Frame: Change in YBOCS from baseline (week 0) to post-treatment (week 6), assessed every 2 weeks. Followup phase data was measured at week 18.
Population: Number Analyzed in Row Differs Due to Missing/Incomplete Data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Transcranial Magnetic Stimulation (TMS) Treatment | Sham-TMS Treatment
Number analyzed (Participants) | 15 | 11
score on a scale
  Week 0 | 23.9 (4.2) | 23.1 (4.1)
  Week 6: number analyzed (Participants) | 10 | 10
  Week 6 | 23.23 (4.4) | 20.6 (5.5)
  Week 18: number analyzed (Participants) | 4 | 4
  Week 18 | 23.5 (3.5) | 17.0 (8.2)

2. Secondary Outcome: Obsessive Compulsive Beliefs as Measured by Obsessive-Compulsive Beliefs Questionnaire (OBQ)
Description: The Obsessive-Compulsive Beliefs Questionnaire (OBQ) is a patient-rated assessment of beliefs considered important in the development and maintenance of obsessive-compulsive disorder (OCD). It contains 44 items ranging from 1 (disagree very much) to 7 (agree very much) across 3-4 thought domains, yielding a total possible score range from 44 to 308. Higher scores indicate more strongly held OCD-related beliefs. We compared the efficacy of TMS to Sham in reducing OCD beliefs over a 6-week period. Efficacy was again compared in the follow-up phase of the study in from week 6 to week 18.
Time Frame: Change in OBQ from baseline (week 0) to post-treatment (week 6), assessed every 2 weeks. Followup phase data was measured at week 18.
Population: Number Analyzed in Row Differs Due to Missing/Incomplete Data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Transcranial Magnetic Stimulation (TMS) Treatment | Sham-TMS Treatment
Number analyzed (Participants) | 15 | 11
score on a scale
  Week 0 | 186.53 (53.29) | 178.91 (33.15)
  Week 6: number analyzed (Participants) | 10 | 10
  Week 6 | 190.60 (63.55) | 180.30 (36.90)
  Week 18: number analyzed (Participants) | 2 | 2
  Week 18 | 220.00 (73.54) | 147.00 (89.10)

3. Secondary Outcome: Total Number of Obsessive Symptoms is Reduced as Measured by Obsessive-Compulsive Inventory Questionnaire (OCI)-Revised
Description: The Obsessive Compulsive Inventory-Revised (OCI-R) is a self-report questionnaire that measures OCD symptoms across 6 sub-scales including washing, checking, neutralizing, obsessing, ordering and hoarding. It contains 18 items ranging from 0 (not at all) to 4 (extremely), yielding a total possible score range from 0 to 72. Higher scores indicate more severe OCD symptoms. We compared the efficacy of TMS to Sham in reducing inventory of obsessive symptoms over a 6-week period. Efficacy was again compared in the follow-up phase of the study in from week 6 to week 18.
Time Frame: Change in OCI from baseline (week 0) to post-treatment (week 6), assessed every 2 weeks. Followup phase data was measured at week 18.
Population: Number Analyzed in Row Differs Due to Missing/Incomplete Data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Transcranial Magnetic Stimulation (TMS) Treatment | Sham-TMS Treatment
Number analyzed (Participants) | 15 | 11
score on a scale
  Week 0 | 26.27 (11.21) | 31.20 (14.05)
  Week 6: number analyzed (Participants) | 10 | 10
  Week 6 | 31.00 (12.32) | 24.70 (11.40)
  Week 18: number analyzed (Participants) | 2 | 2
  Week 18 | 30.50 (10.61) | 15.50 (19.09)

ADVERSE EVENTS:
Time Frame: Adverse event data was assessed during clinician assessments every 2 weeks from baseline (week 0) through week 6 (phase I and phase II), and once more at the end of the 3-month follow-up after phase I (for those not continuing to phase II) or after phase II.
Groups:
- Active Transcranial Magnetic Stimulation (TMS) Treatment (Phase I): In this arm participants received real, active TMS with a standard, water-cooled, figure-8 shaped TMS coil.
  Transcranial Magnetic Stimulation: Transcranial magnetic stimulation uses a rapidly changing magnetic field to induce current in brain tissue non-invasively. It is common procedure in both clinical and research settings, and it has well established guidelines for safe an ethical use which maximize safety for all subjects.
- Sham-TMS Treatment (Phase I): This arm served as the sham/placebo control. In TMS, a sham coil is used to create a sensory experience which is similar to active TMS, but in which the magnetic field is blocked by a metal shield built into the coil.
  Transcranial Magnetic Stimulation: Transcranial magnetic stimulation uses a rapidly changing magnetic field to induce current in brain tissue non-invasively. It is common procedure in both clinical and research settings, and it has well established guidelines for safe an ethical use which maximize safety for all subjects.
- Open-label Active Transcranial Magnetic Stimulation (TMS) Treatment (Phase II): In this arm subjects received real, active TMS with a standard, water-cooled, figure-8 shaped TMS coil.
  Transcranial Magnetic Stimulation: Transcranial magnetic stimulation uses a rapidly changing magnetic field to induce current in brain tissue non-invasively. It is common procedure in both clinical and research settings, and it has well established guidelines for safe an ethical use which maximize safety for all subjects.
Arm/Group | Active Transcranial Magnetic Stimulation (TMS) Treatment (Phase I) | Sham-TMS Treatment (Phase I) | Open-label Active Transcranial Magnetic Stimulation (TMS) Treatment (Phase II)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/11 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/11 | 0/16
Other Adverse Events (participants affected / at risk) | 6/15 | 1/11 | 3/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Transcranial Magnetic Stimulation (TMS) Treatment (Phase I) (N=15) | Sham-TMS Treatment (Phase I) (N=11) | Open-label Active Transcranial Magnetic Stimulation (TMS) Treatment (Phase II) (N=16)
Herniated Disk in Back (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Ear Pain/Pressure (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Minor Car Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
OCD Symptom Worsening (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Flu-Like Symptoms (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Panic Attack (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Sharp Pain in Neck (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Headaches (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Increased Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue After TMS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Increased Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Hypomanic Episode (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Increased Depressive Symptoms (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Nausea Following MRI (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pre-Syncopal Epsiode (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Stomach Bug (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-18): https://cdn.clinicaltrials.gov/large-docs/02/NCT02355002/Prot_SAP_000.pdf